CLINICAL TRIAL: NCT02160509
Title: Telementoring for Emergency Ultrasonography Performed by Emergency Physicians
Brief Title: Telementoring for Emergency Ultrasonography Performed by Emergency Physicians With Low Experience.
Status: Completed | Type: Observational
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Changsun Kim, Professor, Hanyang University
Other Study IDs: 2014-01
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Teleradiology, Ultrasonography
Keywords: real time, ultrasonography, handheld

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- - The patients who undergo ultrasonography in the ED
  Interventions: Device: IPhone based realtime remote ultrasound interpretation

INTERVENTIONS:
Device: IPhone based realtime remote ultrasound interpretation
  Other Names: Application name: cubeview

SUMMARY:
1. Purpose

   * This study aims to evaluate the feasibility of iPhone based telementoring for the ultrasonography.
2. Methods

   * Study Design: Prospective observational study
   * Study Setting: Urban academic ED of tertiary care teaching hospital
   * Study period: July, 2014 ~ December, 2014 (six months)
   * Study participants: Of the patients who need to undergo ultrasonography in the ED, those who are agreed to participate in this study are enrolled.
3. We hypothesize that the iPhone based real time tele-diagnosis by remote expert would not be different from the diagnosis via his/her direct ultrasound examination.

DETAILED DESCRIPTION:
* Teleultrasound system

  1. We already developed the telesystem for viewing the ultrasound examinations performed in the emergency department (ED) by using the iPhone display simultaneously at the out of ED.
  2. Remote mentors can view the patient and examiner's hand holding the ultrasound probe while simultaneously viewing the ultrasound image in the same field of ultrasound display
  3. The examiner and the mentor can communicate with each other.
* Procedures:

  1. The residents perform the ultrasonography and the out of ED expert observe the practice by using the iPhone.
  2. While viewing the practice, the mentor can guide the examiner (resident) to manipulate the probe to get the best ultrasound image.
  3. After finishing the practice, the mentor measures the speed of used mobile network using the application of 'BENCHBEE' and records the predesigned registry.
  4. The registry includes the patients' information, the time and date of examination, the type of mobile network (3G, LTE, WiFi and etc.) and the speed of mobile network, used tele-displayer (iPhone, iPad, iPad mini), used probe, performed body organ (cardiac, lung, Hepatobiliary, vascular, genital organ, appendix and intestine including suspected intussusception), the examiner's level of training and the ultrasound experience of the examiner and the mentor.
  5. The mentor records the patient's diagnosis and the problems during this procedure.
  6. The mentor goes to the patient, perform the ultrasonography directly and confirm the patients' diagnosis.
  7. We will investigate the diagnostic accuracy for iPhone-based tele-ultrasonography comparing these diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* the patients who undergo the emergency physician-performed ultrasonography

Exclusion Criteria:

* the failure of examination due to such as patients' severe obesity, a large amount of gas and etc.
* the patients who refuse to participate in this study.
* the patients who need emergency ultrasonography.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who undergo the ultrasonography in the emergency department
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy by using Receiver Operating Characteristics (area under the curve) | up to 6 months
  Comparing sensitivity and specificity between the iPhone and LCD monitor of the ultrasound machine.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Seung Kang, MD, Study Chair — Emergency Department of Hanyang University
Locations (1):
- Hanyang University guri hospital, Guri-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Kim C, Kang BS, Choi HJ, Lee YJ, Kang GH, Choi WJ, Kwon IH. Nationwide online social networking for cardiovascular care in Korea using Facebook. J Am Med Inform Assoc. 2014 Jan-Feb;21(1):17-22. doi: 10.1136/amiajnl-2012-001465. Epub 2013 May 23. PMID 23703828
- [Background] Park JB, Choi HJ, Lee JH, Kang BS. An assessment of the iPad 2 as a CT teleradiology tool using brain CT with subtle intracranial hemorrhage under conventional illumination. J Digit Imaging. 2013 Aug;26(4):683-90. doi: 10.1007/s10278-013-9580-0. PMID 23404630
- [Background] Lim TH, Choi HJ, Kang BS. Feasibility of dynamic cardiac ultrasound transmission via mobile phone for basic emergency teleconsultation. J Telemed Telecare. 2010;16(5):281-5. doi: 10.1258/jtt.2010.091109. Epub 2010 Jun 24. PMID 20576745
- [Background] Choi HJ, Lee JH, Kang BS. Remote CT reading using an ultramobile PC and web-based remote viewing over a wireless network. J Telemed Telecare. 2012 Jan;18(1):26-31. doi: 10.1258/jtt.2011.110412. Epub 2011 Nov 8. PMID 22067287
- [Background] Biegler N, McBeth PB, Tiruta C, Hamilton DR, Xiao Z, Crawford I, Tevez-Molina M, Miletic N, Ball CG, Pian L, Kirkpatrick AW. The feasibility of nurse practitioner-performed, telementored lung telesonography with remote physician guidance - 'a remote virtual mentor'. Crit Ultrasound J. 2013 Jun 27;5(1):5. doi: 10.1186/2036-7902-5-5. PMID 23805869
- [Background] McBeth P, Crawford I, Tiruta C, Xiao Z, Zhu GQ, Shuster M, Sewell L, Panebianco N, Lautner D, Nicolaou S, Ball CG, Blaivas M, Dente CJ, Wyrzykowski AD, Kirkpatrick AW. Help is in your pocket: the potential accuracy of smartphone- and laptop-based remotely guided resuscitative telesonography. Telemed J E Health. 2013 Dec;19(12):924-30. doi: 10.1089/tmj.2013.0034. Epub 2013 Oct 19. PMID 24138615